CLINICAL TRIAL: NCT00601081
Title: Alterations in the Cytokine Profile of Premature Infants After Human Milk Fortifier
Brief Title: Human Milk Fortifier and Cytokine Profile
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: 27127
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Infant, Very Low Birth Weight
Keywords: Very low birth weight infants; HMF; immune system function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Very low birth weight and preterm infants who will likely receive fortification of breast milk with HMF

SUMMARY:
This is a research study investigating if adding human milk fortifier to a preterm babies breast milk feedings affects the baby's immune system.

DETAILED DESCRIPTION:
In very low birth weight (VLBW) infants and preterm infants human milk fortifier (HMF) is often added to breast milk feedings in order to add extra calories, vitamins, and minerals. It is well known that breast milk feedings are easier to digest and have immune benefits compared to formula feedings. Cytokines, marker of immune function, can be found in blood, stool, and breast milk. This study involves collection of blood and stool samples to monitor cytokines. The purpose of this study is to understand whether human milk fortifier alters infants' cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Infants born weighing less than 1500 grams
* exclusive breast milk feedings with intention to fortify with human milk fortifier

Exclusion Criteria:

* positive blood culture
* history of necrotizing enterocolitis
* significant lung disease at the start of the study

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants hospitalized in the newborn intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Cytokine profile pre and post initiation of HMF | up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert G. Locke, DO, Principal Investigator — Christiana Hospital; Christopher T. Hsu, MD, Principal Investigator — Christiana Hospital
Locations (1):
- Christiana Hospital, Newark, Delaware, United States